CLINICAL TRIAL: NCT02117726
Title: Impact of Various Sedation Regimens on the Incidence of Post-sedation Delirium in Patients Receiving Mechanical Ventilation
Brief Title: Impact of Various Sedation Regimens on the Incidence of Delirium
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Wangchunting, Director, Shandong Provincial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ARDS2014
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Delirium
Keywords: Sedation;; ARDS;; Mechanical ventilation; Hypnotics; Antianxiety Drugs; Causing; Adverse Effects; Therapeutic Use
MeSH Terms: conditions — Delirium | interventions — Dexmedetomidine; Midazolam; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Dexmedetomidine,midazolam (Experimental): Slow injection of 2mg midazolam every minute and watching patients' reaction until attaining the target level of sedation;midazolam was maintained at 0.02~0.1mg/kg/h, for 24 hours.Dexmedetomidine will be added at 0.2~1.4μg/kg/h to maintain sedation.If target sedation level (RASS score) cannot be reached in maximum dose of dexmedetomidine, continuous intravenous infusion of midazolam could be used at 0.02~0.1mg/kg/h, until the target level is reached.
  Interventions: Drug: Dexmedetomidine,midazolam
- Propofol,midazolam (Active Comparator): Slow injection of 2mg midazolam every minute and watching patients' reaction until attaining the target level of sedation;midazolam was maintained at 0.02~0.1mg/kg/h, for 24 hours.Propofol will be added at 0.3~4mg/kg/h to maintain sedation.If target sedation level (RASS score) cannot be reached in maximum dose of propofol, continuous intravenous infusion of midazolam could be used at 0.02~0.1mg/kg/h, until the target level is reached.
  Interventions: Drug: Propofol,midazolam

INTERVENTIONS:
Drug: Dexmedetomidine,midazolam
  Arms: Dexmedetomidine,midazolam
Drug: Propofol,midazolam
  Arms: Propofol,midazolam

SUMMARY:
Sedation drugs that are commonly used in ICU in treatment of ARDS, includes propofol, midazolam and dexmedetomidine . Among these, both dexmedetomidine and propofol have been reported to be used together with midazolam in ICU and the combination of propofol and midazolam is most commonly used, but things follow include a high incidence rate of delirium, But the combination of midazolam and dexmedetomidine may have complementary advantages and could have be a better choice for sedation. In this study, we attempted to observe the effects of two different drug regimens on delirium incidence rates in severe ARDS patients' : midazolam and propofol vs propofol and dexmedetomidine .

ELIGIBILITY:
Inclusion Criteria:

* Subjects willing to give written informed consent.
* Mild, moderate or severe ARDS patients demanding invasive mechanical ventilation.
* Subjects whose expected time of mechanical ventilation is longer than 24 hours.
* Subjects aged between 18 and 70.

Exclusion Criteria:

* Subjects with extremely unstable circulation, whose SBP lower than 90mmHg after volume expansion or pressor agent treatment.
* Subjects with extremely unstable circulation, whose SBP lower than 90mmHg after volume expansion or pressor agent treatment.
* Subjects with heart rates less than 50 beats per minute.
* Subjects with second or third degree atrioventricular block.
* Subjects with serious cerebral injury, severe neurologic disorder (e.g acute stroke, uncontrolled epilepsy and severe dementia) or coma.
* Subjects with acute or severe liver disease (Child-Pugh class C), see attachment 2.
* ARDS patients caused by pulmonary fibrosis or COPD.
* Subjects on all types hemodialysis.
* Subjects with neuromuscular system disease, alcohol withdrawal syndrome or mental disease before entrance of ICU.
* Subjects suspected of narcotic analgesics abusing.
* Subjects needing neuromuscular blocking agents (except intubation).
* Subjects allergic to investigational products or with other contraindication.
* Subjects who are breastfeeding or pregnant
* Subjects participated in other study within 30 days before entrance of ICU

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Incidence rates and duration of delirium | up to 15 days
  Incidence rates and duration of delirium within 14 days after initiation of sedation with dexmedetomidine or propofol
Sedation interruption | up to 5 days
  Eye opening according to the voice orders, eye tracking, clenching fist and nodding are involved in assessment, patients could do 3 of those or more is deemed as conscious and taken in delirium assessment.

SECONDARY OUTCOMES:
Sedation therapy effect | up to 7 days
  The frequency of assessment whose score fall within the target range.
Hospitalized days in ICU | up to 15 days
Death rates | 28 days
  Patients' death rates with a follow-up of 28 days
Incidence rate of patients self-extubation | up to 7 days
Injection speed, total dose and injection of sedatives in different groups. | 7 days
Additional dose of fentanyl and midazolam | up to 7 days
Dosage of diuretic, antiemetic, hypoglycemic, beta-receptor antagonist and vasoactive agents. | up to 15 days
Variation degree of HR, RR, BP and SpO2 | up to 15 days

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - HeNan Tumor Hospital, Zhengzhou, Henan
  - The Second Hospital of Shandong University, Jinan, Shandong
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - Liaocheng Hospital, Liaocheng, Shandong
  - Linyi People's Hospital, Linyi, Shandong
  - Affiliated Hospital of Weifang Medical University, Weifang, Shandong
  - Central Hospital of Zibo, Zibo, Shandong